CLINICAL TRIAL: NCT03660553
Title: Effect of Simplified Insulin Regimen on Glycemic Control and Quality of Life in an Elderly Population With Type 2 Diabetes
Brief Title: Simplified Insulin Regimen for the Elderly
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left University of Miami
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Rajesh Garg, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180541
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Elderly; Insulin treatment; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Subcutaneous Injection (MSI) (Active Comparator): MSI group will receive four insulin injections per day that will include a long acting and a short acting insulin. Short acting insulin will be either insulin aspart or insulin lispro.
  Interventions: Drug: Insulin Glargine; Drug: Insulin Aspart; Drug: Insulin Lispro
- Basal Insulin (BI) (Experimental): BI group will receive only one injection of insulin glargine in the morning.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — 0.40 units/kg body weight
  Arms: Basal Insulin (BI)
Drug: Insulin Glargine — 0.20 units/kg body weight
  Arms: Multiple Subcutaneous Injection (MSI)
Drug: Insulin Aspart — 0.20 units/kg body weight
  Arms: Multiple Subcutaneous Injection (MSI)
Drug: Insulin Lispro — 0.20 units/kg body weight
  Arms: Multiple Subcutaneous Injection (MSI)

SUMMARY:
Basal-bolus insulin therapy, which includes one injection of long acting insulin and three injections of short acting insulin is the most commonly used insulin treatment. However, many older patients find the basal-bolus insulin regimen hard to manage because it involves 4 injections and 4 blood glucose tests each day. It is possible that a simplified treatment that involves one injection of long acting insulin daily and two blood glucose tests daily might be equally effective. This simplified regimen, if effective, would be easier to use and might result in less errors. Therefore, the investigators want to conduct this study to compare using a single daily injection of basal insulin with the usual basal-bolus insulin regimen in elderly patients (age >65 years) with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

-Age >65 years

Exclusion Criteria:

* Unable to provide informed consent
* Enrollment in another research study
* History of hypoglycemia unawareness
* Pregnant women
* Prisoners

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Garg, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Subcutaneous Injection (MSI): Multiple Subcutaneous Injection (MSI) group will receive four insulin injections per day that will include a long acting and a short acting insulin. Short acting insulin will be either insulin aspart or insulin lispro.
  Insulin Glargine: 0.20 units/kg body weight
  Insulin Aspart: 0.20 units/kg body weight
  Insulin Lispro: 0.20 units/kg body weight
- Basal Insulin (BI): Basal Insulin (BI) group will receive only one injection of insulin glargine in the morning.
  Insulin Glargine: 0.40 units/kg body weight
Period: Overall Study
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI)
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HbA1c [Mean (Full Range); unit: %] | 9.9 [7.5 to 12.4] | 7.9 [7 to 8.7] | 8.6 [7 to 12.4]

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c)
Description: The mean HbA1c in the BI group will be compared to the mean HbA1c in the MSI group
Time Frame: 6 months
Measure: Mean (Full Range); unit: percentage of HbA1c
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI)
Number analyzed (Participants) | 3 | 4
percentage of HbA1c | 8.5 [7.4 to 9.7] | 7.8 [7.6 to 8]

2. Secondary Outcome: Incidence of Any Hypoglycemia
Description: Defined as any reported blood glucose (BG) <70 mg/dl will be compared between the two groups
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI)
Number analyzed (Participants) | 3 | 4
participants | 0 | 0

3. Secondary Outcome: Incidence of Severe Hypoglycemia
Description: Any BG <54 mg/dl or patient requiring assistance to recover from hypoglycemia will be compared between 2 groups.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI)
Number analyzed (Participants) | 3 | 4
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Multiple Subcutaneous Injection (MSI) | Basal Insulin (BI)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
This study was terminated and there was insufficient patient data for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03660553/Prot_SAP_001.pdf